CLINICAL TRIAL: NCT06916351
Title: The Effect of Acupressure Applied Before Coronary Angiography on Pain, Anxiety and Vital Signs in Patients
Brief Title: Effect of Acupressure Applied Before CAG on Pain, Anxiety and Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Sarenur Ozen, Nurse, graduate student, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BandirmaOnyediEylul University; Ethics Committee (Other: Approval Number: 2024-89)
Record Dates: First submitted 2025-03-22; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Acupressure; Coronary Angiography and Intervention
Keywords: pain; coronary angiography; anxiety; vital signs; Acupressure; nursing care
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: It is a single-blind, parallel group, pre-test-post-follow-up randomized controlled experimental study.
Who Masked: Participant
Masking Description: The participant does not know which group he/she is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham acupressure (Placebo Comparator): Sham acupressure will be applied to three points parallel to HT7, LI4 and PC6, approximately 1-1.5 cm away from the meridians. To prepare the points for acupressure, these points will be rubbed for approximately 20-30 seconds without applying direct pressure, reducing tissue sensitivity. The researcher will then apply acupressure to these points and symmetrical points using the thumb for three minutes, but will apply less pressure than required levels. Similar to the acupressure group, preparations and acupressure application will take approximately 20 minutes in total for each patient.
  Interventions: Other: Sham acupressure
- Control (No Intervention): Patients in the control group will not receive any intervention and will receive routine treatment and care.
- Acupressure (Experimental): Acupressure will be applied to a total of three points, namely HT7, LI4, and PC6, determined by the researcher with a certificate according to literature and expert opinion before the CAG procedure for the acupressure group. The "cun" measurement unit will be used to determine the points where the application will be made. Before the application, after approximately 20-30 seconds of heating and rubbing without direct pressure on the acupressure points, the researcher will manually press the determined acupressure points with the thumb for 10 seconds to create a depth of 1-1.5 cm. Pressure will be applied to each acupressure point for three consecutive minutes (in the breathing rhythm) without lifting the finger, allowing for two seconds of relaxation. Since the symmetry of the three different points selected on the other extremity will also be applied, a total of 18 minutes of pressure will be applied to each point, with the condition of three minutes.
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure — Acupressure will be applied to a total of three points: the 4th point of the Large Intestine Meridian (LI4-Hegu point) and the 6th point of the pericardial meridian (PC6- Nei Guan point), located three fingers above the wrist.
  Arms: Acupressure
Other: Sham acupressure — Sham acupressure will be applied to three points parallel to HT7, LI4 and PC6, approximately 1-1.5 cm away from the meridians.
  Arms: Sham acupressure

SUMMARY:
This randomized controlled experimental study aimed to determine the effects of acupressure applied before the procedure on pain, anxiety and vital signs in patients who applied to Kocaeli City Hospital Angiography Unit and were to undergo planned radial artery coronary angiography.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted at the Kocaeli City Hospital Angiography Unit to determine the effects of acupressure applied before coronary angiography on pain, anxiety and vital signs of the patients scheduled to undergo coronary angiography. It was conducted at the Kocaeli City Hospital Angiography Unit. The study used a stratified block randomization method and 93 patients who met the inclusion criteria were assigned to two different intervention groups, one of which received acupressure and the other a sham intervention before coronary angiography, and a control group receiving standard care. Data were collected using the 'Personal Information Form', 'State Anxiety Inventory (STAI)', 'Visual Analog Scale (VAS)' and 'Patient Follow-up Form'.

ELIGIBILITY:
Inclusion criteria for the study

* Over 18 years of age,
* Able to understand and speak Turkish,
* Open to communication,
* First time undergoing radial artery coronary angiography,
* Elective patients undergoing planned (non-urgent) coronary angiography,
* Patients who did not undergo stent/balloon intervention during angiography,
* Awake and conscious during coronary intervention (not having taken sedatives (dormicum/fentanyl))
* No deformities or lesions in the areas where acupressure will be applied (hematoma, ecchymosis, etc.)
* Having not taken sedatives or painkillers 5 hours before the angiography,
* No experience with acupressure,
* No history of attending training courses and yoga classes to control stress and anxiety in the last six months
* No diagnosis of anxiety disorder and not receiving medical treatment
* No diagnosis of depression and not receiving medical treatment
* Flat on the back (patients without respiratory distress, etc.),
* Hemodynamically stable (no chest pain or arrhythmia),
* Patients who volunteer to participate in the study,

Exclusion criteria for the study

* Diagnosed with any psychiatric disease
* Previously undergone coronary angiography from the radial or femoral artery
* Chronic pain
* Used opioid medication
* CAG procedure to be performed from the femoral artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale (STAI) | Before acupressure application, 20 minutes after acupressure application (20 minutes after application in the sham acupressure group, 20 min. after the initial measurement in the control group), immediately after the CABG procedure, 2 and 4 hours later
  The State-Trait Anxiety Scale (STAI) is a scale developed by Spielberger et al. in 1970. The STAI determines how an individual feels at a certain moment and under a certain condition. The Turkish adaptation of the STAI was made by Öner and Le Compte in 1983 and the Cronbach alpha coefficient was reported as 0.94 (Öner and Le Compte, 1985). The STAI consists of 20 questions on a four-point Likert type. The statements in the STAI are evaluated as not at all 1 point, a little 2 points, a lot 3 points and completely 4 points. In this section, the statements are divided into direct and reversed. The scale score varies between 20-80 and an increase in the score obtained from the scale indicates an increase in the anxiety level. A score of 0-19 indicates no anxiety, a score of 20-39 indicates mild, a score of 40-59 indicates moderate and a score of 60-79 indicates severe anxiety. It is stated that those who score 60 points and above need professional help.
Visual pain scale for pain assessment | Before acupressure application, 20 minutes after acupressure application (20 minutes after application in the sham acupressure group, 20 min. after the initial measurement in the control group), immediately after the CABG procedure, 2 and 4 hours later
  The scale is a 10 cm vertical or horizontal line on which patients mark their pain, with no pain written on one end and unbearable pain on the other. The distance between where the patient marks their pain and the no pain range is measured and recorded. The scale consists of five parts. Each of the sections is in the range of 2 points. '0' points - no pain, '1-2 points, very mild pain', '3-4 points, mild pain', '5-6 points, moderate pain', '7-8 points, severe pain' means '9-10 points, excruciating pain'.

SECONDARY OUTCOMES:
The blood pressure measurements | Including a total of 5 measurements before the procedure, 20 minutes after the application, immediately after the procedure, 2 hours after the procedure, and 4 hours after the procedure.
  Blood pressure monitoring will be used to evaluate the effects of acupressure, sham and control groups on physiological signs of pain and anxiety. Systolic and diastolic blood pressure measurements are performed by the researcher using the same manual sphygmomanometer instrument. Blood pressure is expressed in "mmHg".
The heart rate measurement | Including a total of 5 measurements before the procedure, 20 minutes after the application, immediately after the procedure, 2 hours after the procedure, and 4 hours after the procedure.
  Heart rate will be used to evaluate the effects of acupressure, sham and control groups on physiological signs of pain and anxiety. Heart rate is measured by the researcher by counting over the radial artery (the untreated artery) for one minute. Heart rate refers to the number of beats per minute.
Respiratory rate | Including a total of 5 measurements before the procedure, 20 minutes after the application, immediately after the procedure, 2 hours after the procedure, and 4 hours after the procedure.
  It will be used to evaluate the effects of breathing, acupressure, sham and control groups on physiological signs of pain and anxiety. Respiratory rate is measured by the researcher by counting the inspiratory and expiratory movements of the chest for one minute. Respiratory rate refers to the number of breaths per minute.
Oxygen saturation | Including a total of 5 measurements before the procedure, 20 minutes after the application, immediately after the procedure, 2 hours after the procedure, and 4 hours after the procedure.
  Oxygen saturation will be used to evaluate the effects of pain and anxiety on hemodynamic parameters in acupressure, sham and control groups. Oxygen saturation was measured by placing a pulse oximeter on the patient's finger, which was used by the researcher to determine the level of oxygen in the blood. The normal reference range for the evaluation of oxygen saturation expressed as SpO2 was accepted as 95-100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No